CLINICAL TRIAL: NCT05301335
Title: Spinal Cord Neuromodulator by SpineX and Scone to Treat Neurogenic Bladder
Brief Title: Spinal COrd NeuromodulaTor by SpIneX and ScoNE to Treat NeurogeniC BladdEr - SCONE "CONTINENCE" Clinical Study
Acronym: CONTINENCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SpineX Inc. (Industry)
Collaborators: Rancho Los Amigos National Rehabilitation Center, Downey, California, United States (Unknown); Atrium Health, Charlotte, North Carolina, United States (Unknown); MedStar National Rehabilitation Network, Washington, District of Columbia, United States (Unknown); University of California, San Diego, California United States (Unknown); Craig Hospital, Englewood, Colorado, United States (Unknown); Columbia University, New York City, New York, United States (Unknown); Institute of Brain and Spine (IBS Hospital), New Delhi, India (Unknown); International Collaboration On Repair Discoveries (ICORD), Vancouver, British Columbia, Canada (Unknown); University of Miami, Miami, United States (Unknown); Mayo Clinic, Rochester, Minnesota, United States (Unknown); Shepherd Center, Atlanta, Georgia, United States (Unknown); Spaulding Rehabilitation Hospital, Charlestown, Massachusetts, United States (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPNX-001
Record Dates: First submitted 2022-03-19; First posted 2022-03-29 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2024-11

CONDITIONS: Neurogenic Bladder; Spinal Cord Injuries (Complete and Incomplete); Stroke; Multiple Sclerosis
MeSH Terms: conditions — Urinary Bladder, Neurogenic; Spinal Cord Injuries; Stroke; Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: The study is designed as a prospective, multicenter, single blind, two-arm randomized sham-controlled clinical study. Subjects will be randomized into a treatment arm and control (sham) arm in a 2:1 ratio.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Therapeutic Arm (Experimental)
  Interventions: Device: SCONE
- Sham Arm (Sham Comparator)
  Interventions: Device: SCONE

INTERVENTIONS:
Device: SCONE — The Spinal COrd NEuromodulation(SCONE) device delivers a sufficient electrical signal non-invasively to activate the neural structures of the spinal cord without cutaneous discomfort. Rather than relying on stimulation of peripheral nerves, SCONE modulates the CNS directly via the spinal cord. Importantly, SCONE is a technique that enables electrical stimulation of the spinal cord without the need for insertion or implantation of stimulating electrodes

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of SCONE neuromodulation therapy after 12 weeks of therapy in comparison to inactive sham control in improving symptoms of Neurogenic Lower Urinary Tract Dysfunction

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 and ≤ 70 years old (male subjects) or ≥ 18 and ≤ 75 years (female subjects) at the time of enrollment/consent.
2. Subject has a diagnosis of NLUTD due to:

   * Chronic, spinal cord injury at C3 to T8 classified as ASIA A-B on the AIS scale OR
   * Chronic, spinal cord injury at C3 to L1 classified as ASIA C-D on the AIS scale OR
   * Multiple sclerosis; OR
   * Stroke
3. Subject has symptoms of urinary urgency (> 50% high urge voids) or increased frequency of micturition/self-catheterization (more than once every 2 hours) or incontinence between voids or catheterizations (> 5/day).
4. Subject has sterile urine or asymptomatic bacteriuria.
5. Subject's score is > 28 on NBSS survey.
6. Subject is at least one year post initial diagnosis of NLUTD at the time of enrollment (consent).
7. Subject's medical condition is stable.
8. Subject has adequate social support network to be able to participate in training and assessment sessions for the duration of the study, at the discretion of the Investigator.
9. Subject has been informed of the nature of the study, can understand the requirements of the study, agrees to participate, and has signed the IRB/REB/EC-approved informed consent.

Exclusion Criteria:

1. Subject relies on an indwelling catheter (urethral or suprapubic) for bladder drainage.
2. Subject has a history of bladder augmentation or continent or incontinent urinary stoma or prior bladder surgery.
3. Subject has congestive heart failure, pulmonary disease necessitating supplemental oxygen use, chronic kidney disease (Stage III or higher), chronic liver disease (Child Pugh class B or C) or poorly controlled diabetes (if diabetic, HbA1c > 8.0 within the preceding 6 months).
4. Subject has a concurrent neurological disease affecting the central nervous system, other than spinal cord injury or multiple sclerosis or stroke.
5. Subject has an implanted central or peripheral neuromodulator.
6. Subject has symptomatic, clinically significant autonomic dysreflexia attacks (characterized by headache and systolic blood pressure greater than 180 mmHg) more than once a week.
7. Subject is dependent on an electromagnetic medical implant (e.g., cardiac pacemaker or implanted drug pump), ventilation support, or other external device.
8. Subject has received intravesical botulinum toxin injection within 12 months preceding enrollment.
9. Subject's BMI is > 35.
10. Subject has history of morphologic bladder outlet obstruction (e.g., due to benign prostatic hyperplasia, urethral stricture and /or bladder neck contracture).
11. Subject has history of frequent symptomatic urinary tract infections, defined as receiving five or more courses of urinary tract infection directed antibiotics within 12 months prior to enrollment.
12. For non catheterizing subjects, post void residual is > 100 mL measured by bladder ultrasound, bladder scanner, or one time catheterization at the time of enrollment
13. For female subjects, history and/or screening responses consistent with pelvic organ prolapse.
14. For non catheterizing male subjects older than 55 years of age, screening responses consistent with benign prostatic hyperplasia.
15. Subjects with significant stress incontinence (> 3 stress incontinence episodes per day), defined as incontinence episodes during physical activity such as cough, sneeze, transfers, and other forms of physical activity.
16. Subject is pregnant or trying to become pregnant; or is nursing.
17. Subject has limited life expectancy or comorbid conditions, social/psychological problems, or cognitive impairments that, in the opinion of the Investigator, will preclude them from participation and completion of study procedures or requirements.
18. Subject has a medical condition or complications related to the use of certain medications that may affect validity of the study as determined by the Investigator.
19. Subject has a medical condition not listed above that may put the subject at risk as determined by the Investigator.
20. Subject is participating in or plans to participate in another research study that may interfere with study endpoints.
21. Subject is known or suspected to be non compliant; and/or subject is unable or unwilling to comply with study requirements.
22. Subject was enrolled after the maximum number of targeted subjects were randomized into the respective disease or UUI group.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Neurogenic Bladder Symptom Score (NBSS) | 12 weeks
  Lower score represents improvements

SECONDARY OUTCOMES:
Urge Urinary Incontinence Episodes | 12 weeks
  Lowered scores represents improvement
Patient Global Improvement Index (PGI-I) | 12 weeks
  Lowered scores represents improvement

CONTACTS AND LOCATIONS:
Locations (12):
- United States (10):
  - Rancho Research Institute, Downey, California
  - UC San Diego Health Systems, San Diego, California
  - Craig Hospital, Denver, Colorado
  - Medstar National Rehab, Washington D.C., District of Columbia
  - University of Miami, Desai Sehti Urology Institute, Miami, Florida
  - Shepherd Centre, Atlanta, Georgia
  - Spaulding Rehabilitation Hospital Cambridge, Cambridge, Massachusetts
  - Mayo Clinic, St. Mary's Campus, Rochester, Minnesota
  - Columbia University Irving Medical Centre, New York, New York
  - Atrium Health, Charlotte, North Carolina
- ICORD Vancouver, Vancouver, British Colombia, Canada
- Insitute of Brain and Spine, New Delhi, New Delhi, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kreydin EI, Abedi A, Morales L, Montero S, Kohli P, Ha N, Chapman D, Abedi A, Ginsberg D, Jann K, Harvey RL, Liu CY. Neural Mechanisms of Poststroke Urinary Incontinence: Results From an fMRI Study. Stroke. 2025 Jun;56(6):1516-1527. doi: 10.1161/STROKEAHA.124.048057. Epub 2025 Apr 10. PMID 40207355
- [Derived] Ha NT, Abedi A, Ojeda LAM, Montero S, Kohli P, Chapman D, Abedi A, Gaburak P, Ginsberg D, Harvey RL, Liu CY, Jann K, Kreydin E. Using Functional Magnetic Resonance Imaging to Detect Differences in Micturition-Related Brain Activity Between Volitional and Involuntary Detrusor Contractions. Neurourol Urodyn. 2025 Feb;44(2):374-381. doi: 10.1002/nau.25655. Epub 2024 Dec 29. PMID 39737577